CLINICAL TRIAL: NCT04129112
Title: Evaluation of Influencing Variables in Awakening Concentration and Concentration at Body Movements of Propofol TCI (Targeted Controlled Infusion) Targeted at the Effector Site
Acronym: TCI
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Federico Linassi, MD, Principal investigator, University of Padova
Other Study IDs: CorMA
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Awareness, Anesthesia
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without body movements: Patient who, under general anesthesia without curare agents, during surgery has no body movements
  Interventions: Drug: We do not modify the normale general anesthesia delivery. We note the concentration of propofol at the effector site of body movementsand awakening
- Patients with body movements: Patient who, under general anesthesia without curare agents, during surgery has any body movements that are no reflexes movements
  Interventions: Drug: We do not modify the normale general anesthesia delivery. We note the concentration of propofol at the effector site of body movementsand awakening

INTERVENTIONS:
Drug: We do not modify the normale general anesthesia delivery. We note the concentration of propofol at the effector site of body movementsand awakening — Propofol in our hospital is routinely delivered by Targeted Controlled Infusion (TCI) pumps. We note the concentration of propofol at the effector site of body movements and awakening

SUMMARY:
Age has been related to awakening propofol concentration at effector site of TCI, but not to the loss of consciousness concentration, neither to the concentration of body movements during surgery, that can be interpreted as a sign of light anesthesia and lead to awareness.

This study aims to determinate the incidence and the propofol TCI concentration at the effector site, in patients undergoing general anaesthesia without NBDs, of any patients body movements, defined as any spontaneous movements (but no reflex movements) during surgery.

DETAILED DESCRIPTION:
Target-Controlled-Infusion (TCI), estimating the effect-size concentration (Ce) of propofol and its elimination time with a computerized system, provides the anaesthesiologist useful information to guide anaesthesia.

Although the correlation between propofol at the effector site at loss of consciousness (Ce LOC) and age is still debated with contrasting results, the correlation between propofol at the effector site at return of consciousness (Ce ROC) and age is well established, and some authors suggested that, due also for age-related changes in both pharmacokinetics and pharmacodynamics of propofol, its dosage should be reduced in elderly patients.

Lowering propofol dosage however, can lead to an higher incidence of awareness during general anaesthesia, even if anaesthesia management is guided by consciousness monitors.

Awareness during anaesthesia has recently been defined not as a binary phenomenon, but as a graded spectra of states and, during general anaesthesia without using neuromuscular blocking drugs (NBDs), body movement on the operating table can be taken as an indication of increasing probability of consciousness or 'light' anaesthesia.

Hence, this study aims to evaluate the impact of age on the concentration at the effector site of propofol-remifentanil anaesthesia administered with TCI pump and without NBDs. Concnetration at the effector site of Propofol at the return of consciousness (CeP ROC) and at any clinical sign of superficialization such as body movements (CeP BM) will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general anesthesia with propofol and remifentanil delivered with TCI infusion pump

Exclusion Criteria:

* neurological or psychiatric or cerebrovascular diseases
* renal insufficiency
* patients unable to understand the information contained in the informed consent form,
* patients with intraoperative hemodynamic instability or
* patients who was delivered curare agents during anaesthesia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: we recruited adult (> 18 years old) undergoing general surgery in Treviso Regional Hospital. We excluded patients with any neurological or psychiatric or cerebrovascular diseases and renal insufficiency in anamnesis, who were unable to understand the information contained in the informed consent form, and patients with intraoperative hemodynamic instability or who was delivered curare agents during anaesthesia.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of body movements in patients undergoing surgery without curare agents | During surgery
  We will note if patients have spontaneous movements during surgery, and calculate the incidence of the phenomenon.

SECONDARY OUTCOMES:
Concentration of propofol at body movements | Patients will be subjected to Sort Portable Mental Status Questionnaire (SPMSQ) before surgery. Other variables are collected during surgery
  We will note the concentration at the effector site of propofol TCI during body movements and compare them to pre-operative and demographical variables (age, weight, height, American Society of Anaesthesiologist physical status classification system (ASA), number of previous general anaesthesia, years of schooling, Sort Portable Mental Status Questionnaire score) and intra-operative variables ( concentration at the effector site of remifentanil at ventilator maladjustment (CeR VM), mean Ce propofol and remifentanil target during maintenance, and maximum, mean and minimum State Entropy (SE) and Response Entropy (RE) values during maintenance).
Concentration of propofol at return of consciousness | Patients will be subjected to Sort Portable Mental Status Questionnaire (SPMSQ) before surgery. Other variables are collected during surgery
  We will note the concentration at the effector site of propofol TCI at awakening and compare them to pre-operative and demographical variables (age, weight, height, American Society of Anaesthesiologist physical status classification system (ASA), number of previous general anaesthesia, years of schooling, Sort Portable Mental Status Questionnaire score) and intra-operative variables ( concentration at the effector site of remifentanil at ventilator maladjustement (CeR VM), mean Ce propofol and remifentanil target during maintenance, and maximum, mean and minimum SE and RE Entropy values during maintenance).

CONTACTS AND LOCATIONS:
Locations (1):
- ULSS 2 Marca Trevigiana, Treviso, Tv, Italy